CLINICAL TRIAL: NCT03841123
Title: Effectiveness of a Dietary Counseling to Prevent Added Sugar and Ultra-processed Foods During the First Year of Life: a Randomized Field Trial
Brief Title: Effectiveness of a Dietary Counseling to Prevent Early Consumption of Added Sugar and Ultra-processed Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Federal University of Bahia (Other); Federal University of Amazonas (Other)
Responsible Party: Principal Investigator, Marcia Regina Vitolo, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UFCSPA-RS
Record Dates: First submitted 2018-12-18; First posted 2019-02-15 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Infant Nutrition Disorders; Feeding Patterns; Health Knowledge, Attitudes, Practice
Keywords: complementary feeding; added sugar; ultra-processed foods; intervention; infants
MeSH Terms: conditions — Infant Nutrition Disorders; Feeding Behavior; Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): At the maternity wards mothers will receive dietary counseling and leaflets as a reminder to prevent the early introduction of added sugar and ultra-processed foods.
  Interventions: Other: Dietary Counseling
- Control (No Intervention): At the maternity wards mothers assigned to control groups will have all the health assistance related to the maternity routine without any interference from the study protocol.

INTERVENTIONS:
Other: Dietary Counseling — The intervention will consist of an individualized, face-to-face, 20 to 30 minute counseling session to mothers by trained health workers who will address healthy eating practices during the first two years of life. A printed, colorful and illustrated material will be used to assist mothers in appropriate food choices, mainly to avoid the introduction of sugar and ultra-processed foods. In addition, they will receive a booklet which addresses the "Ten Steps of Healthy Feeding for children from Birth to Two years of life". The research team will focus on Step2: "Do not give added sugar or foods with added sugar", and Step8:"Do not offer ultra-processed foods as candies and soft drinks". To reinforce the intervention, mothers will receive telephone calls up to the infant reach six months.
  Arms: Intervention

SUMMARY:
The purpose of the study is to prevent the early introduction of added sugar and ultra-processed foods and evaluate the impact on breastfeeding duration, complementary feeding quality, growth and prevalence of caries during the first year of life.

DETAILED DESCRIPTION:
This randomized field trial will be performed at the maternity wards of Friendly Hospitals Initiative in three regions of Brazil: North, Northeast and South. After delivery, mothers who accepted to participate in the study will be randomized into control and intervention groups.It will be performed a weekly block randomization to prevent the contamination of information among mothers of different groups in the same facility. The intervention mothers will be advised not to give added sugar and ultra-processed foods during the first year of life, including a leaflet with colored images as a reminder for mothers. The control group mothers will not receive the study intervention but will be have all the routine health assistance of the maternity. At 6 months and 12 months, mothers of both groups will be visited in their homes and dietary evaluation and anthropometric measurements of their babies will be assessed. At 12 months of age the infants will have dental examinations and hemoglobin concentration through a capillary blood test.

.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age ≥ 37 weeks
* single birth
* Mother with at least 18 years old

Exclusion Criteria:

* Mothers with HIV or HTLV1 positive
* Infants with clinical occurrences or other conditions that prohibit breastfeeding or requires specific dietary treatment.

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 516 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Amount of Added Sugar and ultra-processed foods consumed at 6 months | 6 months
  Information will be obtained through two not consecutive dietary 24 hour recall
Amount of Added Sugar and ultra-processed foods consumed at 12 months | 12 months
  Information will be obtained through two not consecutive dietary 24 hour recall
weight gain pattern at 6 months | 6 months
  Weight at birth and six months will be obtained and the weight gain velocity will be calculated
weight gain pattern at 12 months | 12 months.
  Weight at six months and 12 months will be obtained and the weight gain velocity will be calculated
Number of Participants with dental caries | 12 months
  The dental examination will be performed by dentists
Anemia prevalence | 12 months
  The hemoglobin levels will be obtained by capillary blood tests
Exclusive breastfeeding duration | 6 months
  Proportion of infants from 0-6 months at age who are fed exclusively with breastfeeding
Prevalence of continued breastfeeding at 1 year | 12 months
  Proportion of children 12 months of age who are breastfed

SECONDARY OUTCOMES:
Minimally processed foods, processed foods and total energy intake consumed at 6 months | 6 months
  Information will be obtained through two not consecutive dietary 24 hour recall
Minimally processed foods, processed foods and total energy intake consumed at 12 months | 12 months
  Information will be obtained through two not consecutive dietary 24 hour recall
Offer of added sugar and ultra-processed foods at 6 months | 6 months
  Information will be obtained through a food introduction questionnaire
Offer of added sugar and ultra-processed foods at 12 months | 12 months
  Information will be obtained through a food introduction questionnaire
Proportion of infants from 0-12 months of age who are fed with infant formula, cow's milk and toddler milk | 12 months
  Information will be obtained through a food introduction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marcia R Vitolo, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Federal University of Health Science of Porto Alegre, Porto Alegre, Centro Histórico, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Under Discussion

REFERENCES:
- [Derived] Feldens CA, de Barros Coelho EMR, Vitolo MR, Rogrigues PH, Kramer PF, Peres KG. Effectiveness of a Sugar Consumption Prevention Program in the First Year of Life on the Occurrence of Early Childhood Caries: A Multicentric Randomized Trial in Brazil. Caries Res. 2025;59(3):174-184. doi: 10.1159/000541028. Epub 2024 Oct 30. PMID 39476808
- [Derived] Feldens CA, Heck ABDS, Rodrigues PH, Coelho EMRB, Vitolo MR, Kramer PF. Ankyloglossia and Breastfeeding Duration: A Multicenter Birth Cohort Study. Breastfeed Med. 2024 Jan;19(1):17-25. doi: 10.1089/bfm.2023.0182. PMID 38241126